CLINICAL TRIAL: NCT02305394
Title: Effect of Subanesthetic Dose of Ketamine Combined With Propofol on Cognitive Function in Depressive Patients Undergoing Electroconvulsive Therapy ---a Randomized Control Double-Blind Clinical Trial
Brief Title: Effect of Subanesthetic Dose of Ketamine Combined With Propofol on Cognitive Function in Depressive Patients Undergoing Electroconvulsive Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Min Su, The Department of Anesthesia and Pain Medicine, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CYYYMZ-006
Record Dates: First submitted 2014-11-19; First posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Depressive Symptoms; Impaired Cognition; Electroconvulsive Therapy
Keywords: ketamine; Electroconvulsive Therapy; Cognitive Function
MeSH Terms: conditions — Depression; Cognition Disorders | interventions — Ketamine; Propofol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PK group (ketamine and propofol) (Experimental): propofol 1.5 mg/kg and ketamine 0.3 mg/kg will be administered to participants separately by intravenous infusion.When patients become unconscious, succinylcholine 1 mg/kg (a muscle relaxant) will be administered intravenously. After 1 minute of succinylcholine infused, ECT will be performed with bitemporal electrode placement using a stimulus dose of 1.0-millisecond pulse width, 60-Hz frequency, 6.0-second stimulus duration, and 0.8-A maximal stimulus intensity.
  Interventions: Drug: ketamine and propofol
- P group (propofol group) (Active Comparator): propofol 1.5 mg/kg and normal saline [weight(kg)×0.3÷10]ml will be administered to participants separately by intravenous infusion.When patients become unconscious, succinylcholine 1 mg/kg (a muscle relaxant) will be administered intravenously. After 1 minute of succinylcholine infused, ECT will be performed with bitemporal electrode placement using a stimulus dose of 1.0-millisecond pulse width, 60-Hz frequency, 6.0-second stimulus duration, and 0.8-A maximal stimulus intensity.
  Interventions: Drug: propofol and normal saline

INTERVENTIONS:
Drug: ketamine and propofol — propofol 1.5 mg/kg and ketamine 0.3 mg/kg will be administered to participants separately by intravenous infusion.
  Arms: PK group (ketamine and propofol)
Drug: propofol and normal saline — propofol 1.5 mg/kg and normal saline [weight(kg)×0.3÷10]ml will be administered to participants separately by intravenous infusion.
  Arms: P group (propofol group)

SUMMARY:
Electroconvulsive therapy (ECT) is an effective treatment for depression compared with the current antidepressant agents，but the most important side effect is cognitive dysfunction. The purpose of this study is to determine whether subanesthetic dose of ketamine combined with propofol is superior to propofol anesthesia alone in improving cognitive function in depressive patients undergoing ECT.

DETAILED DESCRIPTION:
Depression is one of the most debilitating and widespread illnesses affecting up to 20% of individuals in their lifetime. However, the current antidepressant agents take weeks to work, and fail to help at least 40% of depressed patients. Electroconvulsive therapy (ECT) is a remarkably effective treatment for depression, but its use is limited by cognitive dysfunction.

As a result, it is becoming a clinical problem which need to be settled urgently. Previous clinical study showed that subanesthetic dose of ketamine could play a role in antidepressant effects with safety and minimal positive psychotic symptoms.The investigators also found that subanesthetic dose of ketamine combined with other anesthetics could improve cognitive function in depressive rats receiving electroconvulsive shock (a model for analogy with ECT). Few clinical researches concerned the effects of subanesthetic dose of ketamine combined with propofol anesthesia on cognitive function in patients after ECT, therefore the investigators conduct this randomized controlled double-blind trial. In this study, cognitive function will be rated by Mini-Mental State examination score.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with moderate or severe depression according to Diagnostic and Statistical Manual of Mental Disorders
2. aged from 18 to 65 years old

Exclusion Criteria:

1. cerebrovascular malformation, arterial aneurysm, hypertension, or glaucoma;
2. classification of American Society of Anesthesiologists physical status score IV or V;
3. complications such as respiratory disease, cardiovascular disease, intracranial hypertension, cerebral vascular disorder;
4. presence of a foreign body such as pacemaker, intracranial electrode, and clips;
5. history of seizures;
6. history of drug abuse;
7. concomitant presence of a mental disorder;
8. pregnancy;
9. history of serious adverse effects related to anesthetics;
10. refusal to consent for the study, or refusal to undergo one single ECT during the first week of therapy.
11. hyperthyreosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State examination score | at 24 hours after the sixth ECT
  Mini-Mental State examination score will be measured at 24 hours after the sixth ECT.

SECONDARY OUTCOMES:
Mini-Mental State examination score | at 24 hours before the first ECT and 24 hours after each ECT, except the sixth ECT.
  Mini-Mental State examination score will be measured at 24 hours before the first ECT and 24 hours after each ECT, except the sixth ECT.
Effects on Antidepression (Hamilton Depression Rating Scale(HDRS) | at 24 hours before the first ECT and 24 hours after each ECT
  Effect on antidepression will be measured by 24-item Hamilton Depression Rating Scale(HDRS)
Seizure Duration and Seizure Energy Index | at 30 seconds after each ECT
  Seizure duration and Seizure energy index will be recorded by the ECT apparatus.
Brief Psychiatric Rating Scale（BPRS） | 60 minutes prior to the first ECT and at 40, 80, 110, and 230 minutes after each ECT
  Brief Psychiatric Rating Scale is related to psychotomimetic side-effect.
Adverse Effects include nausea, vomit, headache, tachycardia and increased blood pressure. | at 40 minutes after each ECT
  Adverse effects include nausea, vomit, headache, tachycardia and increased blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Su Min, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- China,Chongqing The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Machado-Vieira R, Salvadore G, Diazgranados N, Zarate CA Jr. Ketamine and the next generation of antidepressants with a rapid onset of action. Pharmacol Ther. 2009 Aug;123(2):143-50. doi: 10.1016/j.pharmthera.2009.02.010. Epub 2009 May 3. PMID 19397926
- [Background] Garcia LS, Comim CM, Valvassori SS, Reus GZ, Barbosa LM, Andreazza AC, Stertz L, Fries GR, Gavioli EC, Kapczinski F, Quevedo J. Acute administration of ketamine induces antidepressant-like effects in the forced swimming test and increases BDNF levels in the rat hippocampus. Prog Neuropsychopharmacol Biol Psychiatry. 2008 Jan 1;32(1):140-4. doi: 10.1016/j.pnpbp.2007.07.027. Epub 2007 Aug 8. PMID 17884272
- [Background] Berton O, Nestler EJ. New approaches to antidepressant drug discovery: beyond monoamines. Nat Rev Neurosci. 2006 Feb;7(2):137-51. doi: 10.1038/nrn1846. PMID 16429123
- [Background] Pigot M, Andrade C, Loo C. Pharmacological attenuation of electroconvulsive therapy--induced cognitive deficits: theoretical background and clinical findings. J ECT. 2008 Mar;24(1):57-67. doi: 10.1097/YCT.0b013e3181616c14. PMID 18379337
- [Background] aan het Rot M, Collins KA, Murrough JW, Perez AM, Reich DL, Charney DS, Mathew SJ. Safety and efficacy of repeated-dose intravenous ketamine for treatment-resistant depression. Biol Psychiatry. 2010 Jan 15;67(2):139-45. doi: 10.1016/j.biopsych.2009.08.038. PMID 19897179
- [Background] Chen J, Peng LH, Luo J, Liu L, Lv F, Li P, Ao L, Hao XC, Min S. Effects of low-dose ketamine combined with propofol on phosphorylation of AMPA receptor GluR1 subunit and GABAA receptor in hippocampus of stressed rats receiving electroconvulsive shock. J ECT. 2015 Mar;31(1):50-6. doi: 10.1097/YCT.0000000000000148. PMID 24831997
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Price RB, Nock MK, Charney DS, Mathew SJ. Effects of intravenous ketamine on explicit and implicit measures of suicidality in treatment-resistant depression. Biol Psychiatry. 2009 Sep 1;66(5):522-6. doi: 10.1016/j.biopsych.2009.04.029. Epub 2009 Jul 9. PMID 19545857
- [Background] Ibrahim L, Diazgranados N, Luckenbaugh DA, Machado-Vieira R, Baumann J, Mallinger AG, Zarate CA Jr. Rapid decrease in depressive symptoms with an N-methyl-d-aspartate antagonist in ECT-resistant major depression. Prog Neuropsychopharmacol Biol Psychiatry. 2011 Jun 1;35(4):1155-9. doi: 10.1016/j.pnpbp.2011.03.019. Epub 2011 Apr 3. PMID 21466832
- [Background] McDaniel WW, Sahota AK, Vyas BV, Laguerta N, Hategan L, Oswald J. Ketamine appears associated with better word recall than etomidate after a course of 6 electroconvulsive therapies. J ECT. 2006 Jun;22(2):103-6. doi: 10.1097/00124509-200606000-00005. PMID 16801824
- [Background] Krystal AD, Weiner RD, Dean MD, Lindahl VH, Tramontozzi LA 3rd, Falcone G, Coffey CE. Comparison of seizure duration, ictal EEG, and cognitive effects of ketamine and methohexital anesthesia with ECT. J Neuropsychiatry Clin Neurosci. 2003 Winter;15(1):27-34. doi: 10.1176/jnp.15.1.27. PMID 12556568
- [Background] Kranaster L, Kammerer-Ciernioch J, Hoyer C, Sartorius A. Clinically favourable effects of ketamine as an anaesthetic for electroconvulsive therapy: a retrospective study. Eur Arch Psychiatry Clin Neurosci. 2011 Dec;261(8):575-82. doi: 10.1007/s00406-011-0205-7. Epub 2011 Mar 13. PMID 21400226
- [Background] Wang X, Chen Y, Zhou X, Liu F, Zhang T, Zhang C. Effects of propofol and ketamine as combined anesthesia for electroconvulsive therapy in patients with depressive disorder. J ECT. 2012 Jun;28(2):128-32. doi: 10.1097/YCT.0b013e31824d1d02. PMID 22622291
- [Background] Kellner CH, Briggs MC, Pasculli RM, Bryson EO. Antidepressant effect of the first electroconvulsive therapy with ketamine and/or propofol. J ECT. 2013 Jun;29(2):149. doi: 10.1097/YCT.0b013e3182702980. No abstract available. PMID 23703230